CLINICAL TRIAL: NCT04996342
Title: A Cohort Study of Chronic Cardiovascular Diseases in the Department of Cardiology, Peking University First Hospital
Brief Title: A Cohort Study of Chronic Cardiovascular Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jianping LI, Director of Department of Cardiology, Peking University First Hospital
Other Study IDs: CVDcohort
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Diseases; Cohort Studies
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cohort study aims to establish cohorts of patients with chronic cardiovascular disease, including refractory and secondary hypertension, coronary heart disease, atrial fibrillation, ventricular arrhythmias, structural heart disease, pulmonary hypertension, heart failure and rare diseases of the cardiovascular system, and patients with implantations of cardiac pacemaker, in order to dynamically describe the population characteristics, diagnosis and treatment status and long-term prognosis and analyze the factors affecting the choice of treatment plan, long-term management quality and clinical prognosis of these patients.

ELIGIBILITY:
This study includes 9 disease-specific cohorts. The specific inclusion and exclusion criteria are as following:

1. Refractory and secondary hypertension

   Inclusion Criteria:
   * Patients diagnosed as refractory hypertension and/or secondary hypertension
   * Patients willing to accept long-term follow-up and regular return visits

   Exclusion Criteria:
   * Severe diseases of other systems may affecting the life span of patients
2. Coronary heart disease

   Inclusion Criteria:
   * Patients undergoing coronary angiography and interventional therapy in the cath lab
   * Patients undergoing coronary angiography and functional assessment in the cath lab
   * Patients diagnosed as acute myocardial infarction

   Exclusion Criteria:
   * Severe diseases of other systems may affecting the life span of patients
   * Regular return visits not available
3. Atrial fibrillation

   Inclusion Criteria:
   * PAtrial fibrillation diagnosed by electrocardiogram or holter (duration >30 seconds)
   * Patients willing to accept long-term follow-up and regular return visits

   Exclusion Criteria:
   * Severe diseases of other systems may affecting the life span of patients
   * New-onset atrial fibrillation during the perioperative period of major surgery
4. Ventricular arrhythmias

   Inclusion Criteria:
   * Patients diagnosed as ventricular tachycardia, ventricular premature beat
   * Patients willing to accept long-term follow-up and regular return visits

   Exclusion Criteria:
   * Severe diseases of other systems may affecting the life span of patients
   * A transient cause of ventricular arrhythmia was determined by the doctor, and long-term follow-up was not required
5. Cardiac pacemaker implantation

   Inclusion Criteria:
   * Patients with permanent pacemaker implantations due to various causes (including bradycardia pacing, implantable cardioverter defibrillator, cardiac resynchronization therapy, leadless cardiac pacemaker, etc.)
   * Patients willing to accept long-term follow-up and regular return visits

   Exclusion Criteria:
   * Severe diseases of other systems may affecting the life span of patients
6. Structural heart disease

   Inclusion Criteria:
   * Patients diagnosed as structural heart disease, including congenital heart disease and severe valvular disease (moderate and above valvular stenosis or incomplete closure)
   * Patients willing to accept long-term follow-up and regular return visits

   Exclusion Criteria:
   * Severe diseases of other systems may affecting the life span of patients
7. Pulmonary hypertension

   Inclusion Criteria:
   * Patients diagnosed as pulmonary hypertension
   * Patients willing to accept long-term follow-up and regular return visits

   Exclusion Criteria:
   * Severe diseases of other systems may affecting the life span of patients
8. Heart failure

   Inclusion Criteria:
   * Patients diagnosed as heart failure
   * Patients willing to accept long-term follow-up and regular return visits

   Exclusion Criteria:
   * Severe diseases of other systems may affecting the life span of patients
9. Rare diseases of the cardiovascular system

Inclusion Criteria:

* Patients diagnosed as rare diseases in the catalog published by National Health Commission of the People's Republic of China
* Patients willing to accept long-term follow-up and regular return visits

Exclusion Criteria:

* Severe diseases of other systems may affecting the life span of patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the department of Cardiology or outpatient department of Peking University First Hospital will be enrolled if they are aged ≥18 years old, meet the inclusion criteria of each cohort for the 9 specific chronic cardiovascular disease, and need long-term follow-up according to the judgment of doctors after informed consent. Patients will be included in different disease-specific cohorts based on the disease status and treatment, including hypertension, coronary heart disease, arrhythmia (atrial fibrillation, ventricular arrhythmia), pacemaker surgery, structural heart disease, and heart failure, etc. The same patient who meets the inclusion criteria of multiple specific diseases can be entered into different cohorts at the same time. It is expected to enroll 1500 to 2000 patients per year.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 5 year
  Time to the first occurence of Any cause death, myocardial infarction, or Stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Peking University First Hospital, Beijing, Beijing Municipality, China